CLINICAL TRIAL: NCT06298188
Title: Risankizumab in Children With Crohn's Disease (RisaKids): A Multi-center PORTO Group Prospective Study
Brief Title: Risankizumab in Children With Crohn's Disease (RisaKids)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Amit Assa, Pediatric Gastroenterologist, Principal Investigator, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RisaKids
Record Dates: First submitted 2023-10-24; First posted 2024-03-07 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — risankizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Risankizumab (Experimental): Induction regimen: 0,4,8 IV and then every 8 weeks sc
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Risankizumab

SUMMARY:
The goal of this observational study is to to prospectively explore the real life short (12 weeks) and longer term (54 weeks) clinical, biochemical and endoscopic outcomes of risankizumab in pediatric CD.

This is a 1-year prospective multi-center cohort study of children commencing on risankizumab for pediatric CD with 2 years extension for long-term follow-up. The investigators will record clinical manifestations, blood markers and fecal calprotectin, with monitoring for safety signals including infusion and injection site reactions, pyrexia and infections at various intervals as outlined below. The investigators will also include calprotectin monitoring and fecal sample collection for microbiome and serum samples for drug levels. According to available budget, the investigators will also collect fecal and serum samples for metabolome. Samples collection is optional, thus failure of bio-samples collection will not exclude patients from the study.

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of 18 years,
* Patients diagnosed with CD.
* Patients commenced on risankizumab by treating physician (at least one dose), either alone or in combination with any other CD medications, at any stage of the disease.

Exclusion Criteria:

* There will be no exclusion criteria to this study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Co-primary outcomes: Complete remission at end of remission (weeks 12 and week 54) | Through study completion, approximately 3 years
  Co-primary outcomes: Complete remission at end of remission (weeks 12 and week 54) as defined by the fulfilment of all three criteria:
  i. Corticosteroids and enteral nutrition free
  ii. Clinical remission (i.e. PCDAI<10)
  iii. CRP lower than 1 mg/dl (may be substituted by ESR if CRP missing)

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel